CLINICAL TRIAL: NCT00874887
Title: A Clinical Study to Evaluate if Benzalkonium Chloride (BAK) in a Quinolone Eyedrop Reduces the Likelihood of Developing Resistant Organisms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GMA-ZYM-08-001
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-11

CONDITIONS: Anti-biotic Resistance
MeSH Terms: interventions — Moxifloxacin; Gatifloxacin

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Vigamox® (Active Comparator): moxifloxacin 0.5% (m mg/mL), boric acid, sodium chloride, and purified water
  Interventions: Drug: moxifloxacin 0.5% HCI ophthalmic solution
- Zymar® (Active Comparator): gatifloxacin 0.3% (3 mg/mL), benzalkonium chloride 0.005%, edetate disodium; purified water and sodium chloride
  Interventions: Drug: gatifloxacin ophthalmic solution 0.3%

INTERVENTIONS:
Drug: moxifloxacin 0.5% HCI ophthalmic solution — 1 drop in study eye three times a day for 14 days
  Other Names: Vigamox®
  Arms: Vigamox®
Drug: gatifloxacin ophthalmic solution 0.3% — 1 drop in study eye four times a day for 14 days
  Other Names: ZYMAR®
  Arms: Zymar®

SUMMARY:
The purpose of this study is to assess if the presence of BAK in a fluoroquinolone in the study eye affects the development of resistant bacteria on the conjunctiva based upon changes in the surface flora over the course of 2 weeks of topical treatment in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* At least 50 years of age
* In good general health

Exclusion Criteria:

* Any ocular surgery or use of topical antibiotics or antiseptics in either eye within the last 3 months
* Use of topical steroids, or non-steroidal anti inflammatory drugs in either eye within 30 days of Baseline (or anticipated during the study)
* Use of lid scrubs within 7 days of Baseline in either eye (or anticipated use during the study)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Minneapolis, Minnesota, United States
- Saskatoon, Saskatchewan, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Vigamox®: Moxifloxacin 0.5% HCL ophthalmic solution
- Zymar®: Gatifloxacin 0.3% ophthalmic solution
Period: Overall Study
Arm/Group | Vigamox® | Zymar®
Started | 32 | 34
Completed | 32 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vigamox® | Zymar® | Total
Number analyzed (Participants) | 32 | 34 | 66
Age Continuous [Mean (Standard Deviation); unit: years] | 60.3750 (7.8278) | 62.5000 (8.3892) | 61.625 (8.1085)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Strain Resistance of the Conjunctiva as Determined by Minimum Inhibitory Concentration (MIC) at Day 14
Description: Percentage of subjects with strain resistance as determined by Minimum Inhibitory Concentration (MIC) of the conjunctiva (clear membrane covering the white surface of the eye) at day 14. MIC is the lowest concentration of an antimicrobial that inhibits the visible growth of a microorganism after incubation. The MIC cut-off values include: Intermediate is 1 to less than 2; Resistant is greater than or equal to 2.
Time Frame: Day 14
Population: The microbiological (mITT) population consisted of randomized subjects who received study product and had at least one post-baseline microbiological efficacy measure. One patient in the Zymar® group did not have cultures performed at Day 14.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Vigamox® | Zymar®
Number analyzed (Participants) | 32 | 33
Percentage of Subjects | 9.4 | 0

2. Secondary Outcome: Mutant Prevention Concentration (MPC) of the Conjunctiva at Day 14
Description: Mutant Prevention Concentration (MPC) of the conjunctiva (clear membrane covering the white surface of the eye) at day 14. MPC is the lowest drug concentration which prevents growth of any colony of bacteria on the conjunctiva. The MPC outcome measure was not analyzed due to the low number of data points.
Time Frame: Day 14
Population: The microbiological (mITT) population consisted of randomized subjects who received study product and had at least one post-baseline microbiological efficacy measure. Data for this outcome measure were not analyzed due to the low number of data points.
Measure: Number; unit: micrograms per milliliter (ug/mL)
Arm/Group | Vigamox® | Zymar®
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Minimum Inhibitory Concentration 50 (MIC50) at Day 14
Description: The Minimum Inhibitory Concentration 50 (MIC50) is the minimum concentration required to inhibit the growth of 50% of microorganisms. The MIC50 outcome measure was not analyzed due to the low number of data points.
Time Frame: Day 14
Population: as for outcome 2
Measure: Number; unit: micrograms per milliliter (ug/mL)
Arm/Group | Vigamox® | Zymar®
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Minimum Inhibitory Concentration 90 (MIC90) at Day 14
Description: The Minimum Inhibitory Concentration 90 (MIC90) is the minimum concentration required to inhibit the growth of 90% of microorganisms. The MIC90 outcome measure was not analyzed due to the low number of data points.
Time Frame: Day 14
Population: as for outcome 2
Measure: Number; unit: micrograms per milliliter (ug/mL)
Arm/Group | Vigamox® | Zymar®
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Minimum Inhibitory Concentration (MIC) Range at Day 14
Description: MIC range at day 14. MIC is the lowest concentration of an antimicrobial that inhibits the visible growth of a microorganism after incubation. The MIC cut-off values include: Intermediate is 1 to less than 2; Resistant is greater than or equal to 2. The MIC outcome measure was not analyzed due to the low number of data points.
Time Frame: Day 14
Population: as for outcome 2
Measure: Number; unit: micrograms per milliliter (ug/mL)
Arm/Group | Vigamox® | Zymar®
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Vigamox® | Zymar®
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34
Other Adverse Events (participants affected / at risk) | 0/32 | 0/34

LIMITATIONS AND CAVEATS:
Only a small number of resistant species were obtained at the study endpoints. Therefore, some outcome measures were not able to be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo